CLINICAL TRIAL: NCT04373044
Title: A Phase II Randomized Double-Blind Trial of Baricitinib or Placebo Combined With Antiviral Therapy in Patients With Moderate and Severe COVID-19
Brief Title: Baricitinib, Placebo and Antiviral Therapy for the Treatment of Patients With Moderate and Severe COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after the release of results of ACTT-2 (NCT04401579).
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0S-20-3; NCI-2020-02685 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-20-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2020-04-17; First posted 2020-05-04 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: interventions — baricitinib; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm II (placebo, antiviral therapy) (Placebo Comparator): Patients receive placebo PO daily, and standard of care hydroxychloroquine PO TID. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Hydroxychloroquine; Drug: Placebo Administration
- Treatment (baricitinib, antiviral therapy) (Experimental): Patients receive baricitinib PO daily, and standard of care hydroxychloroquine PO TID. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Baricitinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Baricitinib — Given PO
  Other Names: INCB 028050; INCB028050; LY 3009104; LY3009104
  Arms: Treatment (baricitinib, antiviral therapy)
Drug: Hydroxychloroquine — Given PO
Drug: Placebo Administration — Given Po
  Arms: Arm II (placebo, antiviral therapy)

SUMMARY:
This phase II trial studies the effect of baricitinib in combination with antiviral therapy for the treatment of patients with moderate or severe coronavirus disease-2019 (COVID-19). Treatment with antiviral medications such as hydroxychloroquine, lopinavir/ritonavir, and/or remdesivir may act against infection caused by the virus responsible for COVID-19. Baricitinib may reduce lung inflammation. Giving baricitinib in combination with antiviral therapy may reduce the risk of the disease from getting worse and may help prevent the need for being placed on a ventilator should the disease worsen compared to antiviral therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of baricitinib combined with antiviral therapy in participants with COVID-19-related moderate and severe disease in terms of reduction of the proportion of participants requiring invasive mechanical ventilation or dying or requiring anti-IL6 monoclonal antibodies compared to that seen with antiviral alone within 60 days.

SECONDARY OBJECTIVES:

I. To describe the clinical findings in a cohort of symptomatic COVID-19-infected participants.

II. To test whether cytokine signatures predict progression to invasive ventilatory support or death.

III. To describe adverse events (AEs) associated with baricitinib when administered at 4mg in combination with antivirals.

EXPLORATORY OBJECTIVES:

I. Describe the decay in quantitative viral burden from saliva samples collected sequentially under treatment with baricitinib in combination with antivirals.

II. To obtain preliminary data on efficacy and tolerability of baricitinib in combination with antivirals in participants with cancer.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive baricitinib orally (PO) daily, and standard of care hydroxychloroquine PO three times daily (TID). Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive placebo PO daily, and standard of care hydroxychloroquine PO TID. Treatment continues for 14 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for 60 days after enrollment to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Positive polymerase chain reaction (PCR) for severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) in a respiratory tract sample OR positive anti-SARS CoV2 IgM antibody test that is approved by Food and Drug Administration (FDA) or allowed under an emergency use authorization; either result obtained within 5 days prior to study entry
* Cough and/or pneumonia on chest imaging
* Moderate disease with risk factor(s): Peripheral capillary oxygen saturation (SpO2) >= 92% on room air with one of the following risk factors for development of severe disease: age >= 60 years, receiving medication for hypertension, diagnosed diabetes mellitus, known cardiac disease, chronic lung disease, obesity (body mass index [BMI] >= 35 kg/m^2), active malignancy, immunosuppression (receiving biologics or glucocorticoids >= 20 mg/d prednisone equivalent for > 2 weeks)
* Severe disease: SpO2 =< 92% on room air
* Ability to understand and the willingness to sign a written informed consent. Adults not competent to consent will be enrolled with the use of an appropriate legally authorized representative (per California Code, Health and Safety Code - HSC)

  * FDA regulations generally require that the informed consent of a participant be documented by the use of a written consent form approved by the IRB and signed and dated by the participant or the participant's legally authorized representative at the time of consent (21 case form report [CFR] 50.27[a]). In light of COVID-19 infection control measures, the following procedure would satisfy documentation of this requirement if the participant signing the informed consent is in COVID-19 isolation. If the technology is available, electronic methods of obtaining informed consent will be taken. The electronic consent and Health Insurance Portability and Accountability Act (HIPAA) forms will be uploaded and available through REDCap
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 7 days following completion of therapy. NOTE: Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women of child-bearing potential should use highly effective methods of birth control. These are those methods of contraception, alone or in combination, that result in a low failure rate (i.e, less than 1% per year) when used consistently and correctly

Exclusion Criteria:

* Mechanical ventilation, high-flow nasal oxygen, biphasic positive airway pressure (BiPAP)
* Venous thromboembolism within 12 weeks or previously diagnosed thrombophilic conditions or conditions that increase the risk of thrombosis. Individuals with > 1 episode of venous thromboembolism or pulmonary embolism in the past will also be excluded
* Prior receipt of other immunomodulatory drugs (e.g., any JAK inhibitors, immunomodulatory biologics, or other immunomodulatory investigational products) within 14 days prior to enrollment
* Current treatment with probenecid
* Known infection with human immunodeficiency syndrome (HIV), or active infection with hepatitis B or hepatitis C
* Participant with known active or latent tuberculosis infection
* Pregnancy and lactation
* Any serious acute infections or known active or latent tuberculosis

  * All enrolled participants will be screened for latent tuberculosis infection by testing QuantiFERON-TB Gold Plus, but a documented negative test will not be required prior to entry. If a participant is found to have positive QuantiFERON that results after enrollment, baricitinib will be discontinued
* Solid organ transplant recipient
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x upper limit of normal
* Absolute neutrophil count < 1000/mm^3
* Absolute lymphocyte count < 200/mm^3
* Hemoglobin < 8 g/dl
* Estimated glomerular filtration rate (GFR) < 30 mL/min/1.73 m^2
* Any medical condition in the opinion of the investigator that would place the participant at undue high risk for participation in the trial
* Hypersensitivity to the active substance or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring invasive mechanical ventilation or dying | Up to 14 days
  Descriptive statistics, including means, standard deviations, and ranges for continuous variables, as well as percentages and frequencies for categorical variables, will be provided to describe all the clinical findings in a cohort of symptomatic coronavirus disease 2019 (COVID-19)-infected subjects. The collected data will also be graphically presented in boxplots, histograms, and scatter plots. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity, will be made. Group comparisons will be made using either the parametric tests such as t-test and analysis of variance (ANOVA), or the non-parametric statistical method such as Wilcoxon and Kruskal-Wallis tests for continuous variable and Chi-square test for categorical variables. Point estimates, along with the corresponding p-values and 95% confidence intervals will be reported.

SECONDARY OUTCOMES:
Identification of clinical features (vitals signs - body temperature) | Up to 28 days
  Body temperature will be measured in degrees Fahrenheit using an automated thermometer.
Identification of clinical features (vital signs - respiratory rate) | Up to 28 days
  Respiratory rate in times/minute
Identification of clinical features (vital signs - heart rate) | Up to 28 days
  Heart rate in beats/minute
Identification of clinical features (vital signs - blood pressure) | Up to 28 days
  Blood pressure in mmHg
Identification of clinical features (Imaging) | Up to 28 days
  Chest X-ray or pulmonary computed tomography (CT) will be performed
Identification of clinical features (Lab - White Blood Count) | Up to 28 days
  Assessment via standard blood chemistry and metabolic panel
Identification of clinical features (Lab - Absolute Lymphocyte Count) | Up to 28 days
  Assessment via standard blood chemistry and metabolic panel
Identification of clinical features (Lab - Hemoglobin) | Up to 28 days
  Assessment via standard blood chemistry and metabolic panel
Identification of clinical features (Lab - Creatinine) | Up to 28 days
  Assessment via standard blood chemistry and metabolic panel
Identification of biomarkers (C-reactive protein) | Up to 14 days
  CRP is assessed by routinely used determination of CRP.
Identification of biomarkers (Interleukin-6) | Up to 14 days
  IL-6 levels will be assessed using commercial ELISA method
Identification of biomarkers (Tumor Necrosis Factor-alpha) | Up to 14 days
  Tumor Necrosis Factor-alpha as measured in hospital laboratory
Identification of adverse events | Up to 14 days
  Descriptive statistics, including means, standard deviations, and ranges for continuous variables, as well as percentages and frequencies for categorical variables, will be provided to describe all the clinical findings in a cohort of symptomatic COVID-19-infected subjects. The collected data will also be graphically presented in boxplots, histograms, and scatter plots. Investigations for outliers and assumptions for statistical analysis, e.g., normality and homoscedasticity, will be made. Group comparisons will be made using either the parametric tests such as t-test and ANOVA, or the non-parametric statistical method such as Wilcoxon and Kruskal-Wallis tests for continuous variable and Chi-square test for categorical variables. Point estimates, along with the corresponding p-values and 95% confidence intervals will be reported.

OTHER OUTCOMES:
Measurement of COVID19 viral burden | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California